CLINICAL TRIAL: NCT02259842
Title: Safety, Tolerability and Pharmacokinetics of BI 34021 FU2 Oral Drinking Solution in Healthy Male Volunteers (Dose Range: 5 - 500 mg). A Double-blind (Within Dose Groups), Randomised, Placebo-controlled Within Dose Groups, Single Rising Dose Study, Including Re-dosing at 50 mg and 150 mg (Food Effect) and at 100 mg (Two 50 mg Tablets)
Brief Title: Safety, Tolerability and Pharmacokinetics of BI 34021 FU2 Oral Drinking Solution in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1258.1
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Healthy

ARMS (3):
- BI 34021 FU2 solution (Experimental): single rising doses, dose groups 3 and 5 double-dosing (fed and fasted)
  Interventions: Drug: BI 34021 FU2 solution; Other: High fat, high calorie breakfast
- BI 34021 FU2 tablet (Experimental): dose group 4 only
  Interventions: Drug: BI 34021 FU2 tablet
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 34021 FU2 solution
  Arms: BI 34021 FU2 solution
Drug: BI 34021 FU2 tablet — dose group 4 only
  Arms: BI 34021 FU2 tablet
Drug: Placebo
  Arms: Placebo
Other: High fat, high calorie breakfast — only for dose groups 3 and 5
  Arms: BI 34021 FU2 solution

SUMMARY:
Evaluation of safety, tolerability and PK of single rising oral doses of BI 34021 FU2 in healthy male volunteers; comparison of 100 mg drinking solution vs. tablet, assessment of food effect by re-dosing at 50 mg and 150 mg

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests
2. Age ≥21 and Age ≤50 years
3. BMI ≥18.5 and BMI ≤29.9 kg/m2 (Body Mass Index)
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

1. Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
2. Any evidence of a clinically relevant concomitant disease
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
4. Surgery of the gastrointestinal tract (except appendectomy)
5. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
6. History of relevant orthostatic hypotension, fainting spells or blackouts
7. Chronic or relevant acute infections
8. History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
9. Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
10. Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
11. Participation in another trial with an investigational drug within two months prior to administration or during the trial
12. Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
13. Inability to refrain from smoking on trial days
14. Alcohol abuse (more than 60 g/day)
15. Drug abuse
16. Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
17. Excessive physical activities (within one week prior to administration or during the trial)
18. Any laboratory value outside the reference range that is of clinical relevance
19. Inability to comply with dietary regimen of trial site
20. A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
21. A history of additional risk factors for Torsade des Pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
22. Not willing to use adequate contraception (condom use plus another form of contraception e.g. spermicide, oral contraceptive taken by female partner, sterilisation, intrauterine device (IUD) during the whole study period from the time of the first intake of study drug until three months after the last intake

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2008-03; Primary Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with clinically significant findings on physical examination | up to 10 days after last drug administration
Number of participants with clinically significant findings in vital signs | up to 10 days after last drug administration
  blood pressure (BP), pulse rate (PR) respiratory rate (RR), oral body temperature, orthostatic test
Number of participants with clinically significant findings in 12-lead electrocardiogram (ECG) | up to 10 days after last drug administration
Number of participants with clinically significant findings in laboratory tests | up to 10 days after last drug administration
Number of participants with clinically significant findings in safety markers | up to 10 days after last drug administration
  laboratory results for kidney and liver function
Number of participants with adverse events | up to 10 days after last drug administration
Assessment of tolerability by investigator on a 4-point scale | up to 10 days after last drug administration

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma) | up to 72 hours after last drug administration
tmax (time from dosing to maximum measured concentration) | up to 72 hours after last drug administration
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 72 hours after last drug administration
%AUCtz-∞ (the percentage of the AUC0-∞ that is obtained by extrapolation) | up to 72 hours after last drug administration
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 72 hours after last drug administration
AUC0-2h (area under the concentration-time curve of the analytes in plasma over the time interval 0 to 2 hours after drug administration) | up to 2 hours after last drug administration
λz (terminal rate constant in plasma) | up to 72 hours after last drug administration
t1/2 (terminal half-life of the analyte in plasma) | up to 72 hours after last drug administration
MRTp.o. (mean residence time of the analyte in the body after p.o. administration) | up to 72 hours after last drug administration
CL/F (total/apparent clearance of the analyte in plasma after extravascular administration) | up to 72 hours after last drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | up to 72 hours after last drug administration
Aet1-t2 (amount of analyte eliminated in urine from the time point t1 to time point t2) | up to 48 hours after last drug administration
fet1-t2 (fraction of analyte eliminated in urine from time point t1 to time point t2) | up to 48 hours after last drug administration
CLR,t1-t2 (renal clearance of the analyte from the time point t1 until the time point t2) | up to 48 hours after last drug administration